CLINICAL TRIAL: NCT01083953
Title: Optimal End-Tidal Concentration of Sevoflurane and Desflurane for Removal of Supreme Laryngeal Mask Airway in Anaesthetized Adults
Brief Title: Optimal End-Tidal (ET) Sevoflurane and Desflurane Concentration for Extubation of Supreme Laryngeal Mask Airway (LMA) in Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Malaya (Other)
Collaborators: Malaysian Society of Anaesthesiologists (Other)
Responsible Party: Principal Investigator, Cindy Thomas Joseph, doctor, University of Malaya
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: supreme sevo vs des
Record Dates: First submitted 2010-03-08; First posted 2010-03-10 (Estimated); Last update posted 2015-12-03 (Estimated); Status verified 2015-12

CONDITIONS: Airway Complications
Keywords: end tidal concentration
MeSH Terms: interventions — Sevoflurane; Desflurane

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sevoflurane (Experimental): 1 arm will receive sevoflurane at varying concentrations at which extubation is attempted according to the Dixon up and down method
  Interventions: Drug: Sevoflurane
- Desflurane (Experimental): 1 arm will receive desflurane at varying end tidal concentration at which extubation will be attempted according to Dixon up and down method
  Interventions: Drug: Desflurane

INTERVENTIONS:
Drug: Sevoflurane — Comparing the optimal end-tidal concentration sevoflurane and desflurane for LMA extubation
  Arms: Sevoflurane
Drug: Desflurane — Comparing the optimal end-tidal concentration sevoflurane and desflurane for LMA extubation
  Arms: Desflurane

SUMMARY:
The purpose of this study is to determine the optimal volatile anaesthetic (sevoflurane and desflurane) to remove a Supreme LMA in adults in which there is minimal airway response.

Null hypothesis: there is no significant difference between the optimal end tidal concentration of sevoflurane and desflurane for Supreme LMA removal.

DETAILED DESCRIPTION:
The manufactures' instructions for removal of the LMA recommend waiting until protective reflexes have returned. However, the appropriate timing for removal remains controversial. A more frequent incidence of airway hyperreactivity and complications has been reported by some studies when the LMA was removed in the awake state versus the anesthetized state. Techniques that reduce the time from LMA removal to the return of protective airway reflexes would minimize the risk of aspiration, contamination, or airway obstruction.

With increasingly common use of Supreme LMA in anaesthetic practice, a safe and suitable depth for removal of the Supreme LMA requires research.

Thus the determination of the optimal end-tidal concentration of commonly used volatile agents ie. Sevoflurane and Desflurane for Supreme LMA removal requires research, both for patient safety and minimising anaesthetic costs in dealing with airway complications.

ELIGIBILITY:
Inclusion Criteria:

1. ASA 1-2 patients
2. Age 18 - 49 years old
3. Elective surgery of short duration ( < 2 hours ) which require local anaesthetic infiltration

Exclusion Criteria:

1. Upper respiratory tract symptoms in the previous 10 days
2. Risk of gastric oesophageal reflux or regurgitation
3. Known or predicted difficult airway
4. Poor dentition with high risk of damage
5. BMI > 30 kg/m2
6. Refusing to participate

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 54 (Actual)
Dates: Start 2009-11; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Optimal end tidal concentration of sevoflurane/ desflurane | 6 months

SECONDARY OUTCOMES:
presence of airway response | 10 mins after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Cindy Thomas Joseph, Principal Investigator — Department of Anaesthesiology, UMMC
Locations (1):
- University Malaya Medical Centre, Kuala Lumpur, Kuala Lumpur, Malaysia